CLINICAL TRIAL: NCT06137170
Title: Real-world Sequence of Systemic Therapies and Outcomes in Patients With Metastatic Colorectal Cancer Receiving 3rd and 4th Line of Treatment.
Brief Title: A Real-World Study to Learn More About the Order of Different Treatments and Their Effects in People With Metastatic Colorectal Cancer Receiving Their Third and Fourth Line of Treatment
Acronym: RegoSeq
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22581
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAS±BEV-R: Eligible patients who started with trifluridine/tipiracil +/- bevacizumab (TAS+/-Bev) first, followed by regorafenib (R), without other therapies in-between.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- R-TAS±BEV: Eligible patients who started with regorafenib first, followed by TAS+/-Bev without other therapies in-between.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Follow clinical administration.

SUMMARY:
This is an observational study in which data already collected from people with metastatic colorectal cancer will be studied.

Metastatic colorectal cancer (mCRC) is a cancer of the colon (large bowel) or the rectum (lowest part of the bowel just before the anus). Cancer is considered metastatic if it spreads to other parts of the body.

The study drug, regorafenib, is already approved for doctors to prescribe to people with mCRC. It is an anti-cancer drug that blocks several proteins, called enzymes, which are involved in the growth of cancer. Other approved treatments for mCRC include TAS and bevacizumab. The combination of the anti-cancer drugs trifluridine and tipiracil is called TAS. Both TAS and bevacizumab prevent cancer cells from growing and multiplying.

Some studies have shown that people with mCRC who took TAS along with bevacizumab, lived longer than when TAS was taken alone. This may be especially beneficial for patients who have tried other treatments before. However, there is limited knowledge about how and in which order these drugs are given.

To better understand the impact of the order of taking regorafenib and TAS, with or without bevacizumab, more knowledge is needed about how well these treatments work in people with mCRC in European countries.

The main purpose of this study is to learn more about the effects of treatment in people with mCRC who have already received regorafenib and TAS, with or without bevacizumab, one after the other (also called sequential treatment) in a different order.

To do this, researchers will collect the following information:

* how long participants received sequential treatment for mCRC
* number of participants receiving further treatment for mCRC after the sequential treatment
* number and type of further treatments for mCRC
* how long did participants live (also called overall survival).

The data will come from the participants' information stored in health records from 4 centers in 3 European countries including France, Italy, and Spain. The data will be from people with mCRC who started sequential treatment between January 2013 and December 2022 or until the most recent date that allows researchers to assess the participants' health for at least 3 months.

In this study, only available data from routine care are collected. No visits or tests will be required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at diagnosis of mCRC
* Histologically confirmed diagnosis of mCRC
* Received sequential treatment with regorafenib followed by TAS with or without Bevacizumab (R-TAS±BEV, without other therapies in-between) and vice versa (TAS±BEV -R without other therapies in-between) from January 1, 2013 to December 31, 2022 (inclusion period), or the latest available date that allows at least 3 months of follow-up
* Have at least 6 months of available data before index date (baseline period) and at least 3 months of follow-up data

Exclusion Criteria:

* Patients who had a diagnosis of any other primary cancer (including gastrointestinal stromal tumors (GIST) and hepatocellular carcinoma (HCC)) except non-melanoma skin cancers during baseline
* Patients involved in clinical trials during the study period

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective cohort study of patients aged ≥18 years at the diagnosis of mCRC in real world clinical practice who received sequential treatment with regorafenib followed by TAS (with or without Bevacizumab, R-TAS±BEV) and vice versa (TAS±BEV-R) from January 1, 2019 to December 31, 2022 (inclusion period), or the latest available date that allows at least 3 months of follow-up, at multiple clinical centers in France, Italy, and Spain. The study will use longitudinal patients and clinical data recorded at the centers.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Duration of sequential treatment (DoT) | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
Proportion of patients receiving subsequent therapies following sequential treatment during all available follow up after end of sequential treatment | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
Number and type of subsequent therapies | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
Proportion of patients using myelopoiesis supporting therapy | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
Overall Survival (OS) | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up

SECONDARY OUTCOMES:
Descriptive analysis of demographic characteristics | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
ECOG at index (the closest measurement before index date) | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
  Descriptive analysis of clinical characteristics: Descriptive statistics will be calculated. Categorical variables will be summarized using frequency (number of patients [N]) and percentage (%) of total study persons observed in each group. Continuous and count variables will be presented as the mean, standard deviation (SD) and median. As relevant, continuous variables will also be categorized into intervals.
Location of primary cancer: left colon, right colon, rectum | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
  Descriptive analysis of clinical characteristics: Descriptive statistics will be calculated. Categorical variables will be summarized using frequency (number of patients [N]) and percentage (%) of total study persons observed in each group. Continuous and count variables will be presented as the mean, standard deviation (SD) and median. As relevant, continuous variables will also be categorized into intervals.
TNM stage at diagnosis | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
  Descriptive analysis of clinical characteristics: Descriptive statistics will be calculated. Categorical variables will be summarized using frequency (number of patients [N]) and percentage (%) of total study persons observed in each group. Continuous and count variables will be presented as the mean, standard deviation (SD) and median. As relevant, continuous variables will also be categorized into intervals.
Metastasis location: lung, hepatic, other sites | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
  Descriptive analysis of clinical characteristics: Descriptive statistics will be calculated. Categorical variables will be summarized using frequency (number of patients [N]) and percentage (%) of total study persons observed in each group. Continuous and count variables will be presented as the mean, standard deviation (SD) and median. As relevant, continuous variables will also be categorized into intervals.
Molecular diagnostics status | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
  Descriptive analysis of clinical characteristics: Descriptive statistics will be calculated. Categorical variables will be summarized using frequency (number of patients [N]) and percentage (%) of total study persons observed in each group. Continuous and count variables will be presented as the mean, standard deviation (SD) and median. As relevant, continuous variables will also be categorized into intervals.
Regorafenib dose at starting treatment and changes during treatment | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
  Descriptive analysis of clinical characteristics: Descriptive statistics will be calculated. Categorical variables will be summarized using frequency (number of patients [N]) and percentage (%) of total study persons observed in each group. Continuous and count variables will be presented as the mean, standard deviation (SD) and median. As relevant, continuous variables will also be categorized into intervals.
Biomarkers: KRAS, NRAS & BRAF and MMR/MSI | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
Proportion of patients in the sequential treatment groups who received myelopoiesis supporting therapy, differentiating between prophylactic and for therapeutic purpose | Retrospective analysis between January 1, 2013 and December 31, 2022 or the latest available date that allows at least 3 months follow-up
  Myelopoiesis supporting therapy including blood / blood cell transfusions, hematopoietic growth factors, e.g., granulocyte colony stimulating factor and erythropoiesis-stimulating agents.

CONTACTS AND LOCATIONS:
Locations (3):
- Many Locations, Multiple Locations, France
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Spain

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.